CLINICAL TRIAL: NCT02530827
Title: Influence of Lipid-lowering Drugs in Patients Seropositive for HIV With Lipodystrophy in Resting Energy Expenditure and Total Energy Expenditure
Brief Title: Energy Expenditure of People Living With HIV/AIDS
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAAE 01848612.1.0000.5440
Record Dates: First submitted 2015-08-04; First posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: HIV/AIDS; HIV Lipodystrophy Syndrome
Keywords: energy expenditure; doubly labeled water; accelerometer; HIV; lipodystrophy syndrome.
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV-Associated Lipodystrophy Syndrome | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Fibric Acids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- LIPO-HIPO-: HIV-seropositive without lipodystrophy and no use of lipid-lowering drugs.
- LIPO+HIPO-: HIV-seropositive with lipodystrophy and no use of lipid-lowering drugs.
- LIPO+HIPO+: HIV-seropositive with lipodystrophy and use of lipid-lowering drugs.
  Interventions: Drug: use of lipid-lowering drugs.

INTERVENTIONS:
Drug: use of lipid-lowering drugs. — The patients shoud be in use of a lipid-lowering drugs previouly, at least one month before of the begining of the study.
  Other Names: statins and fibrates
  Groups: LIPO+HIPO+

SUMMARY:
Background: Several studies have reported increased resting energy expenditure (REE) in people living with HIV/AIDS possibly due to changes in body composition that occurs in HIV lipodystrophy syndrome.

The aim of this study was to evaluate the influence of the use of lipid-lowering drugs in resting energy expenditure (REE) and total energy expenditure (TEE) in patients seropositive for HIV in treatment of lipodystrophy.

DETAILED DESCRIPTION:
REE was measured by indirect calorimetry.

TEE was measured by doubly labeled water (DLW) technique and an activity monitor based on accelerometry (AM).

ELIGIBILITY:
Inclusion Criteria:

* Use of antiretroviral therapy for at least 4 months
* A cluster of differentiation 4 (CD4) T-cell count of >200 cells/mm3
* Use of lipid-lowering drugs for at least 1 month (group HIV-seropositive with lipodystrophy and use of lipid-lowering)

Exclusion Criteria:

* Signs or symptoms of opportunistic infections
* Thyroid disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men previously diagnosed with HIV infection, on antiretroviral therapy.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Total Energy Expenditure (kcal/d) | 14 day
Resting Energy Expenditure (kcal/d) | 1 day

SECONDARY OUTCOMES:
Correlation between doubly labeled water and accelerometer to measure total energy expenditure (ICC, 95% CI) | 14 days